CLINICAL TRIAL: NCT02189382
Title: Evaluation of the Safety and Efficacy of an Oxalate Gel or Negative Control on Dentinal Hypersensitivity
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Procter and Gamble (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2014029
Record Dates: First submitted 2014-07-08; First posted 2014-07-14 (Estimated); Results first posted 2018-08-20 (Actual); Last update posted 2018-08-20 (Actual); Status verified 2018-07

CONDITIONS: Dentin Sensitivity
Keywords: Sensitivity
MeSH Terms: conditions — Dentin Sensitivity; Hypersensitivity | interventions — Water

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Potassium Oxalate Gel (Experimental): Self Applied
  Interventions: Device: Potassium Oxalate
- Water (Other): Self Applied
  Interventions: Other: Water

INTERVENTIONS:
Device: Potassium Oxalate
  Arms: Potassium Oxalate Gel
Other: Water
  Arms: Water

SUMMARY:
This study will compare the safety and effectiveness of a potassium oxalate desensitizer or negative control on dentinal hypersensitivity.

ELIGIBILITY:
Inclusion Criteria:

* be at least 18 years of age;
* provide written informed consent prior to participation and be given a signed copy of the informed consent form;
* complete a confidentiality disclosure agreement;
* be in good general health as determined by the Investigator/designee;
* agree not to participate in any other oral/dental product studies during the course of this study;
* agree to delay any dentistry (including dental prophylaxis) until the study has been completed;
* agree to refrain from the use of any non-study oral hygiene products;
* agree to return for all scheduled visits and follow study procedures; and.
* have at least one tooth with a Schiff sensitivity score of at least 1 in response to air challenge and a Yeaple Probe score of 10-40 in response to tactile challenge

Exclusion Criteria:

* self-reported pregnancy or nursing;
* severe periodontal disease, as characterized by purulent exudate, generalized mobility, and/or severe recession;
* active treatment of periodontitis;
* fixed facial orthodontic appliances;
* a history of kidney stones;
* known allergies to the following ingredients; aqua, glycerin, cellulose gum, dipotassium oxalate, carbomer, sodium hydroxide, sodium benzoate, and potassium sorbate
* any diseases or conditions that might interfere with the safe completion of the study; or
* an inability to undergo any study procedures.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2014-06; Primary Completion 2014-07 (Actual); Study Completion 2014-07 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Silverstone Research Group, Las Vegas, Nevada, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Potassium Oxalate Gel: Self Applied
  Potassium Oxalate
- Water: Self Applied
  Water
Period: Overall Study
Arm/Group | Potassium Oxalate Gel | Water
Started | 35 | 35
Completed | 35 | 35
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Potassium Oxalate Gel | Water | Total
Number analyzed (Participants) | 35 | 35 | 70
Age, Continuous [Mean (Standard Deviation); unit: years] | 34.5 (11.13) | 36.6 (14.25) | 35.6 (12.74)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 20 | 22 | 42
  Male | 15 | 13 | 28
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Ethnicity: Asian Indian | 0 | 1 | 1
  Ethnicity: Asian Oriental | 2 | 1 | 3
  Ethnicity: Black | 10 | 10 | 20
  Ethnicity: Caucasian | 12 | 14 | 26
  Ethnicity: Hispanic | 9 | 6 | 15
  Ethnicity: Multi-Racial | 2 | 3 | 5

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline Air Challenge
Description: The Schiff Sensitivity Scale was assessed for each test tooth via an evaporative air challenge. The examiner recorded the Schiff Index score corresponding to the response to the air challenge. The Schiff Index Sensitivity scale is scored as follows- 0: tooth/subject did not respond to stimulus, 1: tooth/subject responds to stimulus, but does not request discontinuation of stimulus, 2: tooth/subject responds to stimulus and requests discontinuation or moves form stimulus, 3: tooth/subject responds to stimulus, considers stimulus to be painful, and requests discontinuation of the stimulus. The higher the Schiff score, the more sensitive the tooth. The mean change from Baseline was calculated for this measure.
Time Frame: 30 days
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Potassium Oxalate Gel | Water
Number analyzed (Participants) | 35 | 35
units on a scale | -1.200 (0.677) | -0.086 (0.284)

2. Secondary Outcome: Change From Baseline in Tactile Threshold
Description: Tactile Threshold was measured using a Yeaple probe. Testing was performed beginning at 10 g. The examiner recorded tactile scores for responding teeth. After treatment, testing began at 10 g and increase by 10 g to a maximum of 50 g. The higher the tactile threshold, the less sensitive the tooth. Each successive challenge increased until a "yes" response was repeated. If a second "yes" was not obtained, the force setting was increased to the next step and continued until a force was found which elicited two consecutive "yes" responses and was recorded as the threshold on the Tactile Sensitivity Score form. The mean change from Baseline was calculated for this measure.
Time Frame: 30 days
Measure: Mean (Standard Deviation); unit: Grams (g)
Arm/Group | Potassium Oxalate Gel | Water
Number analyzed (Participants) | 35 | 35
Grams (g) | 16.857 (12.312) | 0.286 (2.956)

ADVERSE EVENTS:
Time Frame: 30 Days
Arm/Group | Potassium Oxalate Gel | Water
All-Cause Mortality (participants affected / at risk) | 0/35 | 0/35
Serious Adverse Events (participants affected / at risk) | 0/35 | 0/35
Other Adverse Events (participants affected / at risk) | 0/35 | 0/35

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Written consent from sponsor.